CLINICAL TRIAL: NCT05527392
Title: Assessing the Effect of Virtual Navigation Interventions to Improve Health Insurance Literacy and Decrease Financial Burden: A Childhood Cancer Survivor Study Randomized Trial (HINTII)
Brief Title: Virtual Health Insurance Navigation Pilot Program for Childhood Survivors (HINTII)
Acronym: HINTII
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elyse Park, PhD, Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000176
Record Dates: First submitted 2022-05-31; First posted 2022-09-02 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Childhood Cancer Survivors
Keywords: Health Insurance; Survivorship

STUDY DESIGN:
Intervention Model Description: Enhanced Usual Care HINT Synchronous Intervention Group HINT Asynchronous Intervention Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HINT Synchronous Intervention Group (HINT-S) (Experimental): a virtual, synchronous version of the 5 HINT-S navigator sessions + HINT booklet
  Interventions: Behavioral: Health Insurance Navigation Tools Program
- HINT Asynchronous Intervention Group (HINT-A) (Experimental): a prerecorded, asynchronous version of the 5 HINT-S navigator sessions + HINT booklet
  Interventions: Behavioral: Health Insurance Navigation Tools Program
- Enhanced Usual Care (No Intervention): HINT Booklet

INTERVENTIONS:
Behavioral: Health Insurance Navigation Tools Program — The program will be delivered via videoconferencing by a navigator over approximately a 3-month period and will consist of 5 sessions. The navigation intervention sessions will be as follows: Section 1- Insurance Plan Basics; Section 2- Your Plan in Relation to Policy; Section 3- Navigating Your Plan and Overcoming Obstacles; Section 4- Managing Care Costs; 5-Understanding Your Medical Bills.
  Arms: HINT Asynchronous Intervention Group (HINT-A); HINT Synchronous Intervention Group (HINT-S)

SUMMARY:
The investigators are conducting a Type I hybrid effectiveness-implementation trial to assess the effectiveness of HINT-S (synchronous) compared to enhanced usual care (EUC) in promoting health insurance literacy, thus reducing worry, unmet health care needs, and financial consequences due to medical costs to improve care and long-term outcomes of childhood cancer survivors. The investigators will also compare HINT-S to HINT-A (asynchronous), a prerecorded, asynchronous version of the 5 HINT-S navigator sessions.

DETAILED DESCRIPTION:
The present study seeks to evaluate a health insurance navigation program with childhood cancer survivors recruited from the Long-Term Follow-Up (LTFU) Cohort. Childhood cancer survivors face health challenges throughout their lives that require monitoring and ongoing care. This is compounded by the tendency among childhood survivors to have higher rates of underinsurance, unmet healthcare needs, and burdensome costs related to care. These burdensome costs also contribute to underutilization of care among survivors. Dr. Park and her colleagues published findings that suggested LTFU survivors had difficulty in understanding how to use their insurance, and often experienced financial-related distress. Understanding and navigating insurance benefits in the current landscape is crucial for cancer survivors to obtain and utilize the health care that they need. With this in mind, the study investigators propose to evaluate the effectiveness of an insurance navigation intervention with LTFU participants, delivered in a synchronous and asynchronous modality.

The navigation intervention will be delivered by a health insurance navigator via HIPAA-compliant videoconferencing for the synchronous group (HINT-S) and will be delivered via pre-recorded video session for the asynchronous group HINT-A). Participants will be randomized into either the two navigation intervention arms (HINT-S and HINT-A; approximately 234 per intervention arm), or the enhanced usual care arm (approximately 52 for control arm). The sample size per arm was chosen to enable evaluation of feasibility and acceptability goals, as well as to explore meaningful differences in the outcomes. To assess the proposed primary and secondary outcomes, all trial participants will complete a baseline and 6-month and 12-month post-program follow-up survey.

ELIGIBILITY:
Inclusion Criteria:

* are 18 years or older at time of enrollment
* are able to give informed consent
* have access to a smartphone, computer, or tablet with internet access
* have US based health insurance
* current LTFU cohort participants
* having access to the CCSS patient portal.

Exclusion Criteria:

* Participants from the pilot trial will not be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Health Insurance Literacy from baseline to 6 months. | 6 months follow up
  Change in Health Insurance Literacy, measured with the validated survey (Health Insurance Literacy scale; HIL), will be compared between groups. The HIL is a 16-item measure of participants' self-reported confidence in understanding of terms (e.g., deductible, co-payments, co-insurance) and confidence in knowing how to do health insurance-related activity (e.g. figuring out co-payments, finding an in-network doctor). Items are rated on a 4-point Likert scale with a total scale score ranging from 16-64; higher scores denote lower literacy.

SECONDARY OUTCOMES:
Change in Health Insurance Literacy from baseline to 12 months. | 12 months follow up
  Change in Health Insurance Literacy, measured with the validated survey (Health Insurance Literacy scale; HIL), will be compared over time between groups. The HIL is a 16-item measure of participants' self-reported confidence in understanding of terms (e.g., deductible, co-payments, co-insurance) and confidence in knowing how to do health insurance-related activity (e.g. figuring out co-payments, finding an in-network doctor). Items are rated on a 4-point Likert scale with a total scale score ranging from 16-64; higher scores denote lower literacy.
Change in self-reported financial hardship from baseline to 12 months. | 12 months follow up
  Change in self-reported financial hardship across time will be compared between groups and measured using 3 scales that tap into 3 domains of financial hardship: a) Behavioral, which assesses unmet health care needs due to health care costs in the past year with 8 yes/no items; more yes scores = more hardship; b) Psychological, which assess worry due to health care costs in the past year with 6-items measured on a 5 point likert; higher score reflects greater worry; c) Material, which assesses the financial consequences of health care cost in the past year with 8 yes/no items; more yes scores = more hardship.
Change in annual out-of-pocket costs from baseline to 12 months. | 12 months follow up
  Change in the dollar amount of out-of-pocket annual costs will be compared over time between groups.
Change in the number of Health Care Visits and Procedures (health care utilization) from baseline to 12 months. | 12 months follow up
  Change in patients healthcare utilization across time will be compared over time between groups.
  Health care utilization will be assessed with 11 items which ask patients to report yes/no to health care visits (e.g., any primary care visits in the past year, usual place of care, receipt of annual vaccinations. A greater number of Yes responses reflects more healthcare use.

CONTACTS AND LOCATIONS:
Overall Officials: Elyse R Park, Ph.D., MPH, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Robison LL, Hudson MM. Survivors of childhood and adolescent cancer: life-long risks and responsibilities. Nat Rev Cancer. 2014 Jan;14(1):61-70. doi: 10.1038/nrc3634. Epub 2013 Dec 5. PMID 24304873
- [Background] Friedman DL, Whitton J, Leisenring W, Mertens AC, Hammond S, Stovall M, Donaldson SS, Meadows AT, Robison LL, Neglia JP. Subsequent neoplasms in 5-year survivors of childhood cancer: the Childhood Cancer Survivor Study. J Natl Cancer Inst. 2010 Jul 21;102(14):1083-95. doi: 10.1093/jnci/djq238. Epub 2010 Jul 15. PMID 20634481
- [Background] Reulen RC, Frobisher C, Winter DL, Kelly J, Lancashire ER, Stiller CA, Pritchard-Jones K, Jenkinson HC, Hawkins MM; British Childhood Cancer Survivor Study Steering Group. Long-term risks of subsequent primary neoplasms among survivors of childhood cancer. JAMA. 2011 Jun 8;305(22):2311-9. doi: 10.1001/jama.2011.747. PMID 21642683
- [Background] Olsen JH, Moller T, Anderson H, Langmark F, Sankila R, Tryggvadottir L, Winther JF, Rechnitzer C, Jonmundsson G, Christensen J, Garwicz S. Lifelong cancer incidence in 47,697 patients treated for childhood cancer in the Nordic countries. J Natl Cancer Inst. 2009 Jun 3;101(11):806-13. doi: 10.1093/jnci/djp104. Epub 2009 May 26. PMID 19470947
- [Background] Mulrooney DA, Yeazel MW, Kawashima T, Mertens AC, Mitby P, Stovall M, Donaldson SS, Green DM, Sklar CA, Robison LL, Leisenring WM. Cardiac outcomes in a cohort of adult survivors of childhood and adolescent cancer: retrospective analysis of the Childhood Cancer Survivor Study cohort. BMJ. 2009 Dec 8;339:b4606. doi: 10.1136/bmj.b4606. PMID 19996459
- [Background] Lipshultz SE, Adams MJ, Colan SD, Constine LS, Herman EH, Hsu DT, Hudson MM, Kremer LC, Landy DC, Miller TL, Oeffinger KC, Rosenthal DN, Sable CA, Sallan SE, Singh GK, Steinberger J, Cochran TR, Wilkinson JD; American Heart Association Congenital Heart Defects Committee of the Council on Cardiovascular Disease in the Young, Council on Basic Cardiovascular Sciences, Council on Cardiovascular and Stroke Nursing, Council on Cardiovascular Radiolo. Long-term cardiovascular toxicity in children, adolescents, and young adults who receive cancer therapy: pathophysiology, course, monitoring, management, prevention, and research directions: a scientific statement from the American Heart Association. Circulation. 2013 Oct 22;128(17):1927-95. doi: 10.1161/CIR.0b013e3182a88099. Epub 2013 Sep 30. No abstract available. PMID 24081971
- [Background] van der Pal HJ, van Dalen EC, van Delden E, van Dijk IW, Kok WE, Geskus RB, Sieswerda E, Oldenburger F, Koning CC, van Leeuwen FE, Caron HN, Kremer LC. High risk of symptomatic cardiac events in childhood cancer survivors. J Clin Oncol. 2012 May 1;30(13):1429-37. doi: 10.1200/JCO.2010.33.4730. Epub 2012 Apr 2. PMID 22473161
- [Background] Armstrong GT, Oeffinger KC, Chen Y, Kawashima T, Yasui Y, Leisenring W, Stovall M, Chow EJ, Sklar CA, Mulrooney DA, Mertens AC, Border W, Durand JB, Robison LL, Meacham LR. Modifiable risk factors and major cardiac events among adult survivors of childhood cancer. J Clin Oncol. 2013 Oct 10;31(29):3673-80. doi: 10.1200/JCO.2013.49.3205. Epub 2013 Sep 3. PMID 24002505
- [Background] Green DM, Kawashima T, Stovall M, Leisenring W, Sklar CA, Mertens AC, Donaldson SS, Byrne J, Robison LL. Fertility of male survivors of childhood cancer: a report from the Childhood Cancer Survivor Study. J Clin Oncol. 2010 Jan 10;28(2):332-9. doi: 10.1200/JCO.2009.24.9037. Epub 2009 Nov 30. PMID 19949008
- [Background] Kadan-Lottick NS, Zeltzer LK, Liu Q, Yasui Y, Ellenberg L, Gioia G, Robison LL, Krull KR. Neurocognitive functioning in adult survivors of childhood non-central nervous system cancers. J Natl Cancer Inst. 2010 Jun 16;102(12):881-93. doi: 10.1093/jnci/djq156. Epub 2010 May 10. PMID 20458059
- [Background] Krull KR, Brinkman TM, Li C, Armstrong GT, Ness KK, Srivastava DK, Gurney JG, Kimberg C, Krasin MJ, Pui CH, Robison LL, Hudson MM. Neurocognitive outcomes decades after treatment for childhood acute lymphoblastic leukemia: a report from the St Jude lifetime cohort study. J Clin Oncol. 2013 Dec 10;31(35):4407-15. doi: 10.1200/JCO.2012.48.2315. Epub 2013 Nov 4. PMID 24190124
- [Background] Ness KK, Krull KR, Jones KE, Mulrooney DA, Armstrong GT, Green DM, Chemaitilly W, Smith WA, Wilson CL, Sklar CA, Shelton K, Srivastava DK, Ali S, Robison LL, Hudson MM. Physiologic frailty as a sign of accelerated aging among adult survivors of childhood cancer: a report from the St Jude Lifetime cohort study. J Clin Oncol. 2013 Dec 20;31(36):4496-503. doi: 10.1200/JCO.2013.52.2268. Epub 2013 Nov 18. PMID 24248696
- [Background] Ness KK, Mertens AC, Hudson MM, Wall MM, Leisenring WM, Oeffinger KC, Sklar CA, Robison LL, Gurney JG. Limitations on physical performance and daily activities among long-term survivors of childhood cancer. Ann Intern Med. 2005 Nov 1;143(9):639-47. doi: 10.7326/0003-4819-143-9-200511010-00007. PMID 16263886
- [Background] Langeveld NE, Grootenhuis MA, Voute PA, de Haan RJ, van den Bos C. Quality of life, self-esteem and worries in young adult survivors of childhood cancer. Psychooncology. 2004 Dec;13(12):867-81. doi: 10.1002/pon.800. PMID 15386796
- [Background] Zeltzer LK, Recklitis C, Buchbinder D, Zebrack B, Casillas J, Tsao JC, Lu Q, Krull K. Psychological status in childhood cancer survivors: a report from the Childhood Cancer Survivor Study. J Clin Oncol. 2009 May 10;27(14):2396-404. doi: 10.1200/JCO.2008.21.1433. Epub 2009 Mar 2. PMID 19255309
- [Background] Ness KK, Gurney JG, Zeltzer LK, Leisenring W, Mulrooney DA, Nathan PC, Robison LL, Mertens AC. The impact of limitations in physical, executive, and emotional function on health-related quality of life among adult survivors of childhood cancer: a report from the Childhood Cancer Survivor Study. Arch Phys Med Rehabil. 2008 Jan;89(1):128-36. doi: 10.1016/j.apmr.2007.08.123. PMID 18164342
- [Background] Brinkman TM, Zhu L, Zeltzer LK, Recklitis CJ, Kimberg C, Zhang N, Muriel AC, Stovall M, Srivastava DK, Robison LL, Krull KR. Longitudinal patterns of psychological distress in adult survivors of childhood cancer. Br J Cancer. 2013 Sep 3;109(5):1373-81. doi: 10.1038/bjc.2013.428. Epub 2013 Jul 23. PMID 23880828
- [Background] Oeffinger KC, Mertens AC, Sklar CA, Kawashima T, Hudson MM, Meadows AT, Friedman DL, Marina N, Hobbie W, Kadan-Lottick NS, Schwartz CL, Leisenring W, Robison LL; Childhood Cancer Survivor Study. Chronic health conditions in adult survivors of childhood cancer. N Engl J Med. 2006 Oct 12;355(15):1572-82. doi: 10.1056/NEJMsa060185. PMID 17035650
- [Background] Hijiya N, Hudson MM, Lensing S, Zacher M, Onciu M, Behm FG, Razzouk BI, Ribeiro RC, Rubnitz JE, Sandlund JT, Rivera GK, Evans WE, Relling MV, Pui CH. Cumulative incidence of secondary neoplasms as a first event after childhood acute lymphoblastic leukemia. JAMA. 2007 Mar 21;297(11):1207-15. doi: 10.1001/jama.297.11.1207. PMID 17374815
- [Background] Hudson MM, Ness KK, Gurney JG, Mulrooney DA, Chemaitilly W, Krull KR, Green DM, Armstrong GT, Nottage KA, Jones KE, Sklar CA, Srivastava DK, Robison LL. Clinical ascertainment of health outcomes among adults treated for childhood cancer. JAMA. 2013 Jun 12;309(22):2371-2381. doi: 10.1001/jama.2013.6296. PMID 23757085
- [Background] Armstrong GT, Kawashima T, Leisenring W, Stratton K, Stovall M, Hudson MM, Sklar CA, Robison LL, Oeffinger KC. Aging and risk of severe, disabling, life-threatening, and fatal events in the childhood cancer survivor study. J Clin Oncol. 2014 Apr 20;32(12):1218-27. doi: 10.1200/JCO.2013.51.1055. Epub 2014 Mar 17. PMID 24638000
- [Background] Public Law 111-148, Patient Protection and Affordable Care Act. www.gpo.gov/fdsys/pkg/PLAW-111publ148/pdf/PLAW-111publ148.pdf
- [Background] Mueller EL, Park ER, Davis MM. What the affordable care act means for survivors of pediatric cancer. J Clin Oncol. 2014 Mar 1;32(7):615-7. doi: 10.1200/JCO.2013.52.6467. Epub 2014 Jan 6. No abstract available. PMID 24395862
- [Background] Tolbert J, Nov 06 ADP, 2020. Key Facts about the Uninsured Population. KFF. Published November 6, 2020. Accessed July 23, 2021. https://www.kff.org/uninsured/issue-brief/key-facts-about-the-uninsured-population/
- [Background] Massachusetts Health Care Reform: Six Years Later. KFF. Published May 2, 2012. Accessed July 23, 2021. https://www.kff.org/health-costs/issue-brief/massachusetts-health-care-reform-six-years-later/
- [Background] Nipp RD, ASCO, Conquer Cancer Foundation Congratulate 2015 Grant and Award Recipients. ASCO Connection. Published June 25, 2015. Accessed July 23, 2021. https://connection.asco.org/magazine/features/asco-conquer-cancer-foundation-congratulate-2015-grant-and-award-recipients
- [Background] Buchmueller T, Carey C, Levy HG. Will employers drop health insurance coverage because of the Affordable Care Act? Health Aff (Millwood). 2013 Sep;32(9):1522-30. doi: 10.1377/hlthaff.2013.0526. PMID 24019355
- [Background] Zhao J, Han X, Zheng Z, Banegas MP, Ekwueme DU, Yabroff KR. Is Health Insurance Literacy Associated With Financial Hardship Among Cancer Survivors? Findings From a National Sample in the United States. JNCI Cancer Spectr. 2019 Oct 21;3(4):pkz061. doi: 10.1093/jncics/pkz061. eCollection 2019 Dec. PMID 32337486
- [Background] Housten AJ, Furtado K, Kaphingst KA, Kebodeaux C, McBride T, Cusanno B, Politi MC. Stakeholders' perceptions of ways to support decisions about health insurance marketplace enrollment: a qualitative study. BMC Health Serv Res. 2016 Nov 8;16(1):634. doi: 10.1186/s12913-016-1890-8. PMID 27821121
- [Background] Landier W, Bhatia S, Eshelman DA, Forte KJ, Sweeney T, Hester AL, Darling J, Armstrong FD, Blatt J, Constine LS, Freeman CR, Friedman DL, Green DM, Marina N, Meadows AT, Neglia JP, Oeffinger KC, Robison LL, Ruccione KS, Sklar CA, Hudson MM. Development of risk-based guidelines for pediatric cancer survivors: the Children's Oncology Group Long-Term Follow-Up Guidelines from the Children's Oncology Group Late Effects Committee and Nursing Discipline. J Clin Oncol. 2004 Dec 15;22(24):4979-90. doi: 10.1200/JCO.2004.11.032. Epub 2004 Dec 2. PMID 15576413
- [Background] Long SK, Goin D. Large Racial and Ethnic Differences in Health Insurance Literacy Signal Need for Targeted Education and Outreach 2014. http://hrms.urban.org/briefs/literacy-by-race.html. Accessed Dec 2, 2014.
- [Background] McCormack L, Bann C, Uhrig J, Berkman N, Rudd R. Health Insurance Literacy of Older Adults. Journal of Consumer Affairs. Summer2009 2009;43(2):223-248.
- [Background] Galbraith AA, Sinaiko AD, Soumerai SB, Ross-Degnan D, Dutta-Linn MM, Lieu TA. Some families who purchased health coverage through the Massachusetts Connector wound up with high financial burdens. Health Aff (Millwood). 2013 May;32(5):974-83. doi: 10.1377/hlthaff.2012.0864. Epub 2013 Apr 17. PMID 23595500
- [Background] Blumberg LJ, Long SK, Kenney GM, Goin D. Public Understanding of Basic Health Insurance Concepts on the Eve of Health Reform | Health Reform Monitoring Survey. Accessed July 23, 2021. http://hrms.urban.org/briefs/hrms_literacy.html
- [Background] Keegan TH, Lichtensztajn DY, Kato I, Kent EE, Wu XC, West MM, Hamilton AS, Zebrack B, Bellizzi KM, Smith AW; AYA HOPE Study Collaborative Group. Unmet adolescent and young adult cancer survivors information and service needs: a population-based cancer registry study. J Cancer Surviv. 2012 Sep;6(3):239-50. doi: 10.1007/s11764-012-0219-9. Epub 2012 Mar 29. PMID 22457219
- [Background] Huang IC, Bhakta N, Brinkman TM, Klosky JL, Krull KR, Srivastava D, Hudson MM, Robison LL. Determinants and Consequences of Financial Hardship Among Adult Survivors of Childhood Cancer: A Report From the St. Jude Lifetime Cohort Study. J Natl Cancer Inst. 2019 Feb 1;111(2):189-200. doi: 10.1093/jnci/djy120. PMID 30085213
- [Background] Dee EC, Nipp RD, Muralidhar V, Yu Z, Butler SS, Mahal BA, Nguyen PL, Sanford NN. Financial worry and psychological distress among cancer survivors in the United States, 2013-2018. Support Care Cancer. 2021 Sep;29(9):5523-5535. doi: 10.1007/s00520-021-06084-1. Epub 2021 Mar 16. PMID 33725174
- [Background] Baedke JL, Lindsey LA, James AS, Huang IC, Ness KK, Howell CR, Brinkman TM, Bhakta N, Ehrhardt MJ, Im C, Letsou W, Liu Q, Robison LL, Hudson MM, Yasui Y. Forgoing needed medical care among long-term survivors of childhood cancer: racial/ethnic-insurance disparities. J Cancer Surviv. 2022 Jun;16(3):677-687. doi: 10.1007/s11764-021-01061-3. Epub 2021 May 27. PMID 34046821
- [Background] Nathan PC, Henderson TO, Kirchhoff AC, Park ER, Yabroff KR. Financial Hardship and the Economic Effect of Childhood Cancer Survivorship. J Clin Oncol. 2018 Jul 20;36(21):2198-2205. doi: 10.1200/JCO.2017.76.4431. Epub 2018 Jun 6. PMID 29874136
- [Background] Fair D, Park ER, Nipp RD, Rabin J, Hyland K, Kuhlthau K, Perez GK, Nathan PC, Armstrong GT, Oeffinger KC, Robison LL, Leisenring W, Kirchhoff AC. Material, behavioral, and psychological financial hardship among survivors of childhood cancer in the Childhood Cancer Survivor Study. Cancer. 2021 Sep 1;127(17):3214-3222. doi: 10.1002/cncr.33613. Epub 2021 Jun 1. PMID 34061973
- [Background] Zafar SY. Financial Toxicity of Cancer Care: It's Time to Intervene. J Natl Cancer Inst. 2015 Dec 11;108(5):djv370. doi: 10.1093/jnci/djv370. Print 2016 May. PMID 26657334
- [Background] Tarnasky AM, Tran GN, Nicolla J, Friedman FAP, Wolf S, Troy JD, Sung AD, Shah K, Oury J, Thompson JC, Gagosian B, Pollak KI, Manners I, Zafar SY. Mobile Application to Identify Cancer Treatment-Related Financial Assistance: Results of a Randomized Controlled Trial. JCO Oncol Pract. 2021 Oct;17(10):e1440-e1449. doi: 10.1200/OP.20.00757. Epub 2021 Apr 2. PMID 33797952
- [Background] Khera N, Kumbamu A, Langer SL, Jatoi A, Kamath CC, Mathew E, Zafar YS, Griffin JM. Developing an Educational Intervention to Address Financial Hardship in Cancer Patients. Mayo Clin Proc Innov Qual Outcomes. 2020 Jul 15;4(4):424-433. doi: 10.1016/j.mayocpiqo.2020.04.004. eCollection 2020 Aug. PMID 32793870
- [Background] Watabayashi K, Steelquist J, Overstreet KA, Leahy A, Bradshaw E, Gallagher KD, Balch AJ, Lobb R, Lavell L, Linden H, Ramsey SD, Shankaran V. A Pilot Study of a Comprehensive Financial Navigation Program in Patients With Cancer and Caregivers. J Natl Compr Canc Netw. 2020 Oct 1;18(10):1366-1373. doi: 10.6004/jnccn.2020.7581. Print 2020 Oct. PMID 33022646
- [Background] Hendriks MJ, Harju E, Roser K, Ienca M, Michel G. The long shadow of childhood cancer: a qualitative study on insurance hardship among survivors of childhood cancer. BMC Health Serv Res. 2021 May 25;21(1):503. doi: 10.1186/s12913-021-06543-9. PMID 34034742
- [Background] Sinaiko AD, Ross-Degnan D, Soumerai SB, Lieu T, Galbraith A. The experience of Massachusetts shows that consumers will need help in navigating insurance exchanges. Health Aff (Millwood). 2013 Jan;32(1):78-86. doi: 10.1377/hlthaff.2012.0124. PMID 23297274
- [Background] Centers for Medicare & Medicaid Services (CMS), Department of Health and Human Services (HHS). Patient Protection and Affordable Care Act; Exchange functions: standards for Navigators and non-Navigator assistance personnel; consumer assistance tools and programs of an Exchange and certified application counselors. Final rule. Fed Regist. 2013 Jul 17;78(137):42823-62. PMID 23866380
- [Background] Phillips CE, Rothstein JD, Beaver K, Sherman BJ, Freund KM, Battaglia TA. Patient navigation to increase mammography screening among inner city women. J Gen Intern Med. 2011 Feb;26(2):123-9. doi: 10.1007/s11606-010-1527-2. Epub 2010 Oct 8. PMID 20931294
- [Background] Percac-Lima S, Grant RW, Green AR, Ashburner JM, Gamba G, Oo S, Richter JM, Atlas SJ. A culturally tailored navigator program for colorectal cancer screening in a community health center: a randomized, controlled trial. J Gen Intern Med. 2009 Feb;24(2):211-7. doi: 10.1007/s11606-008-0864-x. PMID 19067085
- [Background] Pollitz K. Data Note: Limited Navigator Funding for Federal Marketplace States. KFF. Published October 13, 2020. Accessed July 20, 2021. https://www.kff.org/private-insurance/issue-brief/data-note-further-reductions-in-navigator-funding-for-federal-marketplace-states/
- [Background] Marketplace Enrollment Tops 12 Million For 2021; Largest-Ever Funding For Navigators | Health Affairs Blog. Accessed July 22, 2021. https://www.healthaffairs.org/do/10.1377/hblog20210422.65513/full/
- [Background] Pratt-Chapman M, Simon MA, Patterson AK, Risendal BC, Patierno S. Survivorship navigation outcome measures: a report from the ACS patient navigation working group on survivorship navigation. Cancer. 2011 Aug;117(15 Suppl):3575-84. doi: 10.1002/cncr.26261. PMID 21780092
- [Background] Park ER, Li FP, Liu Y, Emmons KM, Ablin A, Robison LL, Mertens AC; Childhood Cancer Survivor Study. Health insurance coverage in survivors of childhood cancer: the Childhood Cancer Survivor Study. J Clin Oncol. 2005 Dec 20;23(36):9187-97. doi: 10.1200/JCO.2005.01.7418. PMID 16361621
- [Background] Park ER, Kirchhoff AC, Zallen JP, Weissman JS, Pajolek H, Mertens AC, Armstrong GT, Robison LL, Donelan K, Recklitis CJ, Diller LR, Kuhlthau KA. Childhood Cancer Survivor Study participants' perceptions and knowledge of health insurance coverage: implications for the Affordable Care Act. J Cancer Surviv. 2012 Sep;6(3):251-9. doi: 10.1007/s11764-012-0225-y. Epub 2012 May 17. PMID 22592507
- [Background] Kirchhoff AC, Kuhlthau K, Pajolek H, Leisenring W, Armstrong GT, Robison LL, Park ER. Employer-sponsored health insurance coverage limitations: results from the Childhood Cancer Survivor Study. Support Care Cancer. 2013 Feb;21(2):377-83. doi: 10.1007/s00520-012-1523-7. Epub 2012 Jun 21. PMID 22717916
- [Background] Park ER, Kirchhoff AC, Perez GK, Leisenring W, Weissman JS, Donelan K, Mertens AC, Reschovsky JD, Armstrong GT, Robison LL, Franklin M, Hyland KA, Diller LR, Recklitis CJ, Kuhlthau KA. Childhood Cancer Survivor Study participants' perceptions and understanding of the Affordable Care Act. J Clin Oncol. 2015 Mar 1;33(7):764-72. doi: 10.1200/JCO.2014.58.0993. Epub 2015 Feb 2. PMID 25646189
- [Background] Kuhlthau KA, Nipp RD, Shui A, Srichankij S, Kirchhoff AC, Galbraith AA, Park ER. Health insurance coverage, care accessibility and affordability for adult survivors of childhood cancer: a cross-sectional study of a nationally representative database. J Cancer Surviv. 2016 Dec;10(6):964-971. doi: 10.1007/s11764-016-0542-7. Epub 2016 Apr 12. PMID 27072683
- [Background] Park ER, Kirchhoff AC, Nipp RD, Donelan K, Leisenring WM, Armstrong GT, Kuhlthau KA. Assessing Health Insurance Coverage Characteristics and Impact on Health Care Cost, Worry, and Access: A Report From the Childhood Cancer Survivor Study. JAMA Intern Med. 2017 Dec 1;177(12):1855-1858. doi: 10.1001/jamainternmed.2017.5047. PMID 28973059
- [Background] Nipp RD, Kirchhoff AC, Fair D, Rabin J, Hyland KA, Kuhlthau K, Perez GK, Robison LL, Armstrong GT, Nathan PC, Oeffinger KC, Leisenring WM, Park ER. Financial Burden in Survivors of Childhood Cancer: A Report From the Childhood Cancer Survivor Study. J Clin Oncol. 2017 Oct 20;35(30):3474-3481. doi: 10.1200/JCO.2016.71.7066. Epub 2017 Aug 17. PMID 28817372
- [Background] Perez GK, Kirchhoff AC, Recklitis C, Krull KR, Kuhlthau KA, Nathan PC, Rabin J, Armstrong GT, Leisenring W, Robison LL, Park ER. Mental health insurance access and utilization among childhood cancer survivors: a report from the childhood cancer survivor study. J Cancer Surviv. 2018 Aug;12(4):528-536. doi: 10.1007/s11764-018-0691-y. Epub 2018 Apr 15. PMID 29658062
- [Background] Galbraith AA, Ross-Degnan D, Soumerai SB, Rosenthal MB, Gay C, Lieu TA. Nearly half of families in high-deductible health plans whose members have chronic conditions face substantial financial burden. Health Aff (Millwood). 2011 Feb;30(2):322-31. doi: 10.1377/hlthaff.2010.0584. PMID 21289354
- [Background] Penfold RB, Kullgren JT, Miroshnik I, Galbraith AA, Hinrichsen VL, Lieu TA. Reliability of a patient survey assessing cost-related changes in health care use among high deductible health plan enrollees. BMC Health Serv Res. 2011 May 27;11:133. doi: 10.1186/1472-6963-11-133. PMID 21619647
- [Background] Wisk LE, Gangnon R, Vanness DJ, Galbraith AA, Mullahy J, Witt WP. Development of a novel, objective measure of health care-related financial burden for U.S. families with children. Health Serv Res. 2014 Dec;49(6):1852-74. doi: 10.1111/1475-6773.12248. Epub 2014 Oct 18. PMID 25328073
- [Background] Galbraith AA, Ross-Degnan D, Soumerai SB, Miroshnik I, Wharam JF, Kleinman K, Lieu TA. High-deductible health plans: are vulnerable families enrolled? Pediatrics. 2009 Apr;123(4):e589-94. doi: 10.1542/peds.2008-1738. PMID 19336350
- [Background] Galbraith AA, Ross-Degnan D, Soumerai SB, Abrams AM, Kleinman K, Rosenthal MB, Wharam JF, Adams AS, Miroshnik I, Lieu TA. Use of well-child visits in high-deductible health plans. Am J Manag Care. 2010 Nov;16(11):833-40. PMID 21348554
- [Background] Lieu TA, Solomon JL, Sabin JE, Kullgren JT, Hinrichsen VL, Galbraith AA. Consumer awareness and strategies among families with high-deductible health plans. J Gen Intern Med. 2010 Mar;25(3):249-54. doi: 10.1007/s11606-009-1184-5. Epub 2009 Dec 22. PMID 20033623
- [Background] Wharam JF, Landon BE, Galbraith AA, Kleinman KP, Soumerai SB, Ross-Degnan D. Emergency department use and subsequent hospitalizations among members of a high-deductible health plan. JAMA. 2007 Mar 14;297(10):1093-102. doi: 10.1001/jama.297.10.1093. PMID 17356030
- [Background] Wharam JF, Galbraith AA, Kleinman KP, Soumerai SB, Ross-Degnan D, Landon BE. Cancer screening before and after switching to a high-deductible health plan. Ann Intern Med. 2008 May 6;148(9):647-55. doi: 10.7326/0003-4819-148-9-200805060-00004. PMID 18458277
- [Background] Emmons KM, Puleo E, Park E, Gritz ER, Butterfield RM, Weeks JC, Mertens A, Li FP. Peer-delivered smoking counseling for childhood cancer survivors increases rate of cessation: the partnership for health study. J Clin Oncol. 2005 Sep 20;23(27):6516-23. doi: 10.1200/JCO.2005.07.048. Epub 2005 Aug 22. PMID 16116148
- [Background] Park ER, Puleo E, Butterfield RM, Zorn M, Mertens AC, Gritz ER, Li FP, Emmons KM. A process evaluation of a telephone-based peer-delivered smoking cessation intervention for adult survivors of childhood cancer: the partnership for health study. Prev Med. 2006 Jun;42(6):435-42. doi: 10.1016/j.ypmed.2006.03.004. Epub 2006 Apr 19. PMID 16626797
- [Background] Park EB, Emmons KM, Malloy NW, Seifer E. A qualitative exploration of health perceptions and behaviors among adult survivors of childhood cancers. J Cancer Educ. 2002 Winter;17(4):211-5. doi: 10.1080/08858190209528840. PMID 12556058
- [Background] Butterfield RM, Park ER, Puleo E, Mertens A, Gritz ER, Li FP, Emmons K. Multiple risk behaviors among smokers in the childhood cancer survivors study cohort. Psychooncology. 2004 Sep;13(9):619-29. doi: 10.1002/pon.764. PMID 15334530
- [Background] Duffey-Lind EC, O'Holleran E, Healey M, Vettese M, Diller L, Park ER. Transitioning to survivorship: a pilot study. J Pediatr Oncol Nurs. 2006 Nov-Dec;23(6):335-43. doi: 10.1177/1043454206293267. PMID 17035624
- [Background] Earle CC, Park ER, Lai B, Weeks JC, Ayanian JZ, Block S. Identifying potential indicators of the quality of end-of-life cancer care from administrative data. J Clin Oncol. 2003 Mar 15;21(6):1133-8. doi: 10.1200/JCO.2003.03.059. PMID 12637481
- [Background] Wescott P.H., Reifler, E. J., Sepucha, K., Park, E. R. Breast cancer treatment decision making: Does the sisterhood of breast cancer transcend culture? Research in the Sociology of Health Care: Health Care Services, Racial and Ethnic Minorities and Underserved Populations 2005; 23.
- [Background] Bober SL, Park ER, Schmookler T, Medeiros Nancarrow C, Diller L. Perceptions of breast cancer risk and cancer screening: a qualitative study of young, female Hodgkin's disease survivors. J Cancer Educ. 2007 Spring;22(1):42-6. doi: 10.1007/BF03174374. PMID 17570808
- [Background] Warner EL, Wu YP, Hacking CC, Wright J, Spraker-Perlman HL, Gardner E, Kirchhoff AC. An Assessment to Inform Pediatric Cancer Provider Development and Delivery of Survivor Care Plans. J Cancer Educ. 2015 Dec;30(4):677-84. doi: 10.1007/s13187-015-0829-9. PMID 25893925
- [Background] Mann K, Wu YP, Pannier ST, Hacking C, Warner EL, Rosen S, Acharya A, Wright J, Gerdy C, Kirchhoff AC. Healthcare provider perspectives on pediatric cancer survivorship care plans: a single institution pilot study. Support Care Cancer. 2021 Feb;29(2):697-706. doi: 10.1007/s00520-020-05522-w. Epub 2020 May 21. PMID 32435970
- [Background] Pannier ST, Mann K, Warner EL, Rosen S, Acharya A, Hacking C, Gerdy C, Wright J, Wu YP, Kirchhoff AC. Survivorship care plan experiences among childhood acute lymphoblastic leukemia patients and their families. BMC Pediatr. 2019 Apr 13;19(1):111. doi: 10.1186/s12887-019-1464-0. PMID 30979365
- [Background] Waters AR, Mann K, Vaca Lopez PL, Kepka D, Wu YP, Kirchhoff AC. HPV Vaccine Experiences and Preferences Among Young Adult Cancer Survivors and Caregivers of Childhood Cancer Survivors. J Cancer Educ. 2022 Oct;37(5):1519-1524. doi: 10.1007/s13187-021-01992-6. Epub 2021 Mar 19. PMID 33740231
- [Background] Balaban RB, Galbraith AA, Burns ME, Vialle-Valentin CE, Larochelle MR, Ross-Degnan D. A Patient Navigator Intervention to Reduce Hospital Readmissions among High-Risk Safety-Net Patients: A Randomized Controlled Trial. J Gen Intern Med. 2015 Jul;30(7):907-15. doi: 10.1007/s11606-015-3185-x. Epub 2015 Jan 24. PMID 25617166
- [Background] Burns ME, Galbraith AA, Ross-Degnan D, Balaban RB. Feasibility and evaluation of a pilot community health worker intervention to reduce hospital readmissions. Int J Qual Health Care. 2014 Aug;26(4):358-65. doi: 10.1093/intqhc/mzu046. Epub 2014 Apr 16. PMID 24744082
- [Background] Donelan K, Mailhot JR, Dutwin D, Barnicle K, Oo SA, Hobrecker K, Percac-Lima S, Chabner BA. Patient perspectives of clinical care and patient navigation in follow-up of abnormal mammography. J Gen Intern Med. 2011 Feb;26(2):116-22. doi: 10.1007/s11606-010-1436-4. Epub 2010 Jul 7. PMID 20607432
- [Background] Kuhlthau KA, Luberto CM, Traeger L, Millstein RA, Perez GK, Lindly OJ, Chad-Friedman E, Proszynski J, Park ER. A Virtual Resiliency Intervention for Parents of Children with Autism: A Randomized Pilot Trial. J Autism Dev Disord. 2020 Jul;50(7):2513-2526. doi: 10.1007/s10803-019-03976-4. PMID 30900195
- [Background] Park ER, Perez GK, Millstein RA, Luberto CM, Traeger L, Proszynski J, Chad-Friedman E, Kuhlthau KA. A Virtual Resiliency Intervention Promoting Resiliency for Parents of Children with Learning and Attentional Disabilities: A Randomized Pilot Trial. Matern Child Health J. 2020 Jan;24(1):39-53. doi: 10.1007/s10995-019-02815-3. PMID 31650412
- [Background] Perez GK, Walsh EA, Quain K, Abramson JS, Park ER. A virtual resiliency program for lymphoma survivors: helping survivors cope with post-treatment challenges. Psychol Health. 2021 Nov;36(11):1352-1367. doi: 10.1080/08870446.2020.1849699. Epub 2020 Nov 28. PMID 33251861
- [Background] Mazurek MO, Stobbe G, Loftin R, Malow BA, Agrawal MM, Tapia M, Hess A, Farmer J, Cheak-Zamora N, Kuhlthau K, Sohl K. ECHO Autism Transition: Enhancing healthcare for adolescents and young adults with autism spectrum disorder. Autism. 2020 Apr;24(3):633-644. doi: 10.1177/1362361319879616. Epub 2019 Oct 3. PMID 31581793
- [Background] Park ER, Sylvia LG, Streck JM, Luberto CM, Stanton AM, Perez GK, Baim M, Bliss CC, Convery MS, Crute S, Denninger JW, Donelan K, Dossett ML, Fava M, Fredriksson S, Fricchione G, George N, Hall DL, Hart BR, Herman J, Hirschberg A, Holt D, Looby SE, Malloy L, Meek J, Mehta DH, Millstein RA, Mizrach H, Rosa K, Slawsby E, Stupinski AC, Traeger L, Vanderkruik R, Vogeli C, Wilhelm S. Launching a resiliency group program to assist frontline clinicians in meeting the challenges of the COVID-19 pandemic: Results of a hospital-based systems trial. Gen Hosp Psychiatry. 2021 Jan-Feb;68:111-112. doi: 10.1016/j.genhosppsych.2020.10.005. Epub 2020 Nov 2. No abstract available. PMID 33229013
- [Background] DeTore N, Shannon A, Hynes S, Herman J, Perlis R, Fava M, Park ER, Sylvia L, Holt DJ. Resilience and levels of emotional distress in healthcare workers during the COVID-19 pandemic. MGH Clinical Research Day. Boston, MA. October 2021.
- [Background] Rigotti NA, Bitton A, Kelley JK, Hoeppner BB, Levy DE, Mort E. Offering population-based tobacco treatment in a healthcare setting: a randomized controlled trial. Am J Prev Med. 2011 Nov;41(5):498-503. doi: 10.1016/j.amepre.2011.07.022. PMID 22011421
- [Background] Rigotti NA, Regan S, Levy DE, Japuntich S, Chang Y, Park ER, Viana JC, Kelley JH, Reyen M, Singer DE. Sustained care intervention and postdischarge smoking cessation among hospitalized adults: a randomized clinical trial. JAMA. 2014 Aug 20;312(7):719-28. doi: 10.1001/jama.2014.9237. PMID 25138333
- [Background] Delahanty LM, Dalton KM, Porneala B, Chang Y, Goldman VM, Levy D, Nathan DM, Wexler DJ. Improving diabetes outcomes through lifestyle change--A randomized controlled trial. Obesity (Silver Spring). 2015 Sep;23(9):1792-9. doi: 10.1002/oby.21172. Epub 2015 Aug 11. PMID 26260043
- [Background] Levy DE, Munshi VN, Ashburner JM, Zai AH, Grant RW, Atlas SJ. Health IT-assisted population-based preventive cancer screening: a cost analysis. Am J Manag Care. 2015 Dec;21(12):885-91. PMID 26671700
- [Background] Celano CM, Healy B, Suarez L, Levy DE, Mastromauro C, Januzzi JL, Huffman JC. Cost-Effectiveness of a Collaborative Care Depression and Anxiety Treatment Program in Patients with Acute Cardiac Illness. Value Health. 2016 Mar-Apr;19(2):185-91. doi: 10.1016/j.jval.2015.12.015. Epub 2016 Feb 6. PMID 27021752
- [Background] Levy DE, Klinger EV, Linder JA, Fleegler EW, Rigotti NA, Park ER, Haas JS. Cost-Effectiveness of a Health System-Based Smoking Cessation Program. Nicotine Tob Res. 2017 Nov 7;19(12):1508-1515. doi: 10.1093/ntr/ntw243. PMID 27639095
- [Background] Delahanty LM, Levy DE, Chang Y, Porneala BC, Goldman V, McCarthy J, Bissett L, Rodriguez AR, Chase B, LaRocca R, Wheeler A, Wexler DJ. Effectiveness of Lifestyle Intervention for Type 2 Diabetes in Primary Care: the REAL HEALTH-Diabetes Randomized Clinical Trial. J Gen Intern Med. 2020 Sep;35(9):2637-2646. doi: 10.1007/s11606-019-05629-9. Epub 2020 Jan 21. PMID 31965526
- [Background] Drouin O, Sato R, Drehmer JE, Nabi-Burza E, Hipple Walters B, Winickoff JP, Levy DE. Cost-effectiveness of a Smoking Cessation Intervention for Parents in Pediatric Primary Care. JAMA Netw Open. 2021 Apr 1;4(4):e213927. doi: 10.1001/jamanetworkopen.2021.3927. PMID 33792730
- [Background] Altice CK, Banegas MP, Tucker-Seeley RD, Yabroff KR. Financial Hardships Experienced by Cancer Survivors: A Systematic Review. J Natl Cancer Inst. 2016 Oct 20;109(2):djw205. doi: 10.1093/jnci/djw205. Print 2017 Feb. PMID 27754926
- [Background] de Souza JA, Yap BJ, Wroblewski K, Blinder V, Araujo FS, Hlubocky FJ, Nicholas LH, O'Connor JM, Brockstein B, Ratain MJ, Daugherty CK, Cella D. Measuring financial toxicity as a clinically relevant patient-reported outcome: The validation of the COmprehensive Score for financial Toxicity (COST). Cancer. 2017 Feb 1;123(3):476-484. doi: 10.1002/cncr.30369. Epub 2016 Oct 7. PMID 27716900
- [Background] Levy H, Meltzer D. What Do We Really Know About Whether Health Insura.pdf. Accessed July 23, 2021. https://web.stanford.edu/~jay/health_class/Readings/Lecture02/levy_meltzer.pdf
- [Background] Aday LA, Andersen R. A framework for the study of access to medical care. Health Serv Res. 1974 Fall;9(3):208-20. PMID 4436074
- [Background] Andersen RM. Revisiting the behavioral model and access to medical care: does it matter? J Health Soc Behav. 1995 Mar;36(1):1-10. PMID 7738325
- [Background] Andersen RM. National health surveys and the behavioral model of health services use. Med Care. 2008 Jul;46(7):647-53. doi: 10.1097/MLR.0b013e31817a835d. PMID 18580382
- [Background] Demographics of Mobile Device Ownership and Adoption in the United States. Pew Research Center: Internet, Science & Tech. Accessed May 28, 2021.
- [Background] https://www.pewresearch.org/fact-tank/2021/07/16/home-broadband-adoption-computer-ownership-vary-by-race-ethnicity-in-the-u-s/
- [Background] Bhatia S, Gibson TM, Ness KK, Liu Q, Oeffinger KC, Krull KR, Nathan PC, Neglia JP, Leisenring W, Yasui Y, Robison LL, Armstrong GT. Childhood cancer survivorship research in minority populations: A position paper from the Childhood Cancer Survivor Study. Cancer. 2016 Aug 1;122(15):2426-39. doi: 10.1002/cncr.30072. Epub 2016 Jun 2. PMID 27253866
- [Background] https://ccss.stjude.org/data-and-analysis/public-access-data-tables.html.
- [Background] https://www.neighborhoodatlas.medicine.wisc.edu/
- [Background] Holahan J, Long S. Health Reform Monitoring Survey, first quarter 2016 [Internet]. Ann Arbor (MI): Inter-university Consortium for Political and Social Research [distributor]; 2017 Apr 28 [cited 2019 Jan 31]. Available from: https://www.icpsr.umich.edu/icpsrweb/HMCA/studies/36744/version/1
- [Background] Sinaiko AD, Hayes M, Kingsdale J, Peltz A, Galbraith AA. Understanding Consumer Experiences and Insurance Outcomes Following Plan Disenrollment in the Nongroup Insurance Market. Med Care Res Rev. 2022 Feb;79(1):36-45. doi: 10.1177/1077558721998910. Epub 2021 Mar 16. PMID 33724071
- [Background] Hero JO, Sinaiko AD, Kingsdale J, Gruver RS, Galbraith AA. Decision-Making Experiences Of Consumers Choosing Individual-Market Health Insurance Plans. Health Aff (Millwood). 2019 Mar;38(3):464-472. doi: 10.1377/hlthaff.2018.05036. PMID 30830810
- [Background] Yabroff KR, Zhao J, Han X, Zheng Z. Prevalence and Correlates of Medical Financial Hardship in the USA. J Gen Intern Med. 2019 Aug;34(8):1494-1502. doi: 10.1007/s11606-019-05002-w. Epub 2019 May 1. PMID 31044413
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Mueller EL, Park ER, Kirchhoff AC, Kuhlthau K, Nathan PC, Perez GK, Rabin J, Hutchinson R, Oeffinger KC, Robison LL, Armstrong GT, Leisenring WM, Donelan K. Insurance, chronic health conditions, and utilization of primary and specialty outpatient services: a Childhood Cancer Survivor Study report. J Cancer Surviv. 2018 Oct;12(5):639-646. doi: 10.1007/s11764-018-0700-1. Epub 2018 Jun 25. PMID 29943170
- [Background] Kurt BA, Nolan VG, Ness KK, Neglia JP, Tersak JM, Hudson MM, Armstrong GT, Hutchinson RJ, Leisenring WM, Oeffinger KC, Robison LL, Arora M. Hospitalization rates among survivors of childhood cancer in the Childhood Cancer Survivor Study cohort. Pediatr Blood Cancer. 2012 Jul 15;59(1):126-32. doi: 10.1002/pbc.24017. Epub 2011 Dec 16. PMID 22180128
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Overview of BLS Wage Data by Area and Occupation : U.S. Bureau of Labor Statistics. Accessed July 22, 2021. https://www.bls.gov/bls/blswage.htm
- [Derived] Park ER, Kirchhoff AC, Mitchell CO, Durieux N, Foor A, Kuhlthau K, Perez GK, Ards L, Alston S, Armstrong GT, Vaca Lopez PL, McDonald A, Nolan VG, Levy DE, Leisenring WM, Galbraith AA, Nathan PC, Vukadinovich C, Cooper CL, Donelan K. Assessing the effect of virtual navigation interventions to improve health insurance literacy and decrease financial burden in cancer survivors: The HINT II study protocol. Contemp Clin Trials. 2025 Jul;154:107952. doi: 10.1016/j.cct.2025.107952. Epub 2025 May 12. PMID 40368025